CLINICAL TRIAL: NCT05190809
Title: Immediate Breast Reconstruction With Hybrid Fat Transfer: Prospective Single-arm Interventional Study
Brief Title: Immediate Breast Reconstruction With Hybrid Fat Transfer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abouqir General Hospital (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abouzaid, Dr. Ahmed Mohamed Abouzaid, Abouqir General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0304743
Record Dates: First submitted 2021-12-21; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Breast Appearance Reconstruction Disproportion
Keywords: Goldilocks Mastectomy; Fat grafting; Breast reconstruction; skin sparing mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Group of female patients who will undergo Goldilocks mastectomy in which they will receive an autologous fat grafting in the remaining breast flaps
  Interventions: Procedure: Goldilocks mastectomy and fat transfer

INTERVENTIONS:
Procedure: Goldilocks mastectomy and fat transfer — Skin sparing mastectomy (Goldilocks mastectomy), then autologous fat grafting in the medial and lateral breast pillars as well as the inferior dermal flap

SUMMARY:
Investigators in this study describe a new perspective for female patients that will undergo skin-sparing mastectomy in which there will be an immediate reconstruction of the mastectomized breast for more satisfactory aesthetic results.

DETAILED DESCRIPTION:
This study introduces a new perspective for women who will undergo mastectomy especially Goldilocks mastectomy in which the investigators do fat grafting to the medial and lateral pillars of the breast as well as the inferior dermal flap in order to have a voluminous remaining breast shape that is close enough in size with the contralateral breast for more aesthetic results and to observe the lipografted tissue reaction after radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Age 20 - 65 years old
* females with unilateral breast malignancy
* candidate for Goldilocks mastectomy procedure

Exclusion Criteria:

* Females with ages beyond the study frame.
* Females refusing to participate
* Fameles that not accepting the liposuction, lipofilling procedure
* Females with contralateral previously operated or mastectomized breast.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Immediate breast reconstruction and equalizing the operated breast cup size with the no-operated breast cup size | 6 months follow up post-surgical
  fat grafting to the Goldilocks mastectomy flaps to have the mastectomized breast cup size to be aesthetically close to the contralateral non-operated breast cup size, also 5 point Likert scale was used to evaluate the patient satisfaction

SECONDARY OUTCOMES:
Evaluate the skin changes and the trophic effect of radiotherapy on the fat grafted tissue | through the radiotherapy course and 1 month after
  observe and evaluate the skin changes to the skin flaps of the mastectomy side after radiotherapy and evaluate if the fat grafted tissue can resist the trophic effect of radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Abouqir General Hospital, Alexandria, Egypt